CLINICAL TRIAL: NCT07375498
Title: Phase 1 Clinical Study of the Safety and Pharmacokinetics of Rescue Liposome in Healthy Adult Participants
Brief Title: Safety and Pharmacokinetics of Rescue Liposome in Healthy Adults
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cristália Produtos Químicos Farmacêuticos Ltda. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRT115
Record Dates: First submitted 2026-01-13; First posted 2026-01-29 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Healthy Adult; Overdose Antidote
Keywords: pharmacokinetic; safety

STUDY DESIGN:
Intervention Model Description: The innovative investigational drug is a liposomal dispersion that functions as an effective detoxifying agent by sequestering circulating intoxicants and removing excess levels from the bloodstream. This mechanism supports the reversal of clinical signs of overdose and the prevention of tissue damage. Given its novel nature, the proposed study aims to evaluate the safety and tolerability of the product in healthy participants using a cohort-based dose-escalation design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CRIS115 treatment (Experimental): Injectable liposomal dispersion with a concentration of 22.08 mg/mL
  Interventions: Drug: liposome dispersion

INTERVENTIONS:
Drug: liposome dispersion — liposome rescue

SUMMARY:
This is a Phase 1 study to assess the safety and tolerability of the liposomal product in healthy participants.

DETAILED DESCRIPTION:
This is a Phase 1 clinical trial consisting of a dose-escalation and dose-expansion study to evaluate the safety, clinical tolerability, and pharmacokinetics of the intravenous liposomal dispersion product in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent form (ICF).
* Age ≥ 18 years and ≤ 30 years.
* Body mass index (BMI) between 18.5 and 30.0 kg/m².
* Be able to complete the study in accordance with the protocol requirements.
* Health status: no mental disorders and no history of diseases of the cardiovascular, nervous, respiratory, digestive, urinary, or endocrine systems, and no metabolic abnormalities.
* Willingness to use effective contraception.

Exclusion Criteria:

* Having donated blood within 6 months prior to admission or having experienced significant blood loss (> 450 mL).
* Having participated in any clinical trial involving investigational drugs within 6 months prior to admission in the study.
* Positive test for hepatitis B, hepatitis C, syphilis, and/or HIV.
* Safety laboratory values outside the normal reference range.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-08-20 (Estimated); Primary Completion 2026-12-20 (Estimated); Study Completion 2027-02-20 (Estimated)

PRIMARY OUTCOMES:
Safety: Number of Treatment Related Adverse Events | From enrollment to the end of treatment at 2 weeks.
  The severity/intensity (grade 1 to grade 5) of adverse events will be assessed by the investigator as "unlikely," "possibly," or "probably" related to the investigational drug. An adverse event will be considered causally related to the use of the investigational drug when the causality assessment was "probable" or "possible."
Safety: Number of Clinically Significant (CS) Changes in Physical Examination. | From enrollment to the end of treatment at 2 weeks.
  A complete physical examination includes assessments of selected body systems, at the investigator's discretion, but covers at least the cardiovascular, pulmonary, and neurological systems.
  Examination results will be documented in the eCRF as normal, abnormal without clinical significance (CNS), or abnormal with clinical significance (CS). Post-dose physical examination findings classified as abnormal CS will be reported as adverse events (AEs).

SECONDARY OUTCOMES:
Cmax | From time 0 (time of dosing) to 10,080 minutes after dose (concentration measured at timepoints pre-dose and 0; 5; 10; 15; 20; 40; 50; 60; 70; 90 120; 240; 360; 540; 720; 1,440; 2,160; 2,880 and 10,080 minutes post-dose).
  The Maximal Plasma Concentration (Cmax) after a single dose of liposome in fasting conditions.
AUC | From time 0 (time of dosing) to 10,080 minutes after dose (concentration measured at timepoints pre-dose and 0; 5; 10; 15; 20; 40; 50; 60; 70; 90 120; 240; 360; 540; 720; 1,440; 2,160; 2,880 and 10,080 minutes post-dose).
  AUC will be determined by evaluating the pharmacokinetic profile, in which the liposome in the blood will be quantified.
T1/2(z) | From time 0 (time of dosing) to 10,080 minutes after dose (concentration measured at timepoints pre-dose and 0; 5; 10; 15; 20; 40; 50; 60; 70; 90 120; 240; 360; 540; 720; 1,440; 2,160; 2,880 and 10,080 minutes post-dose).
  Plasma half-life associated with the terminal elimination phase (T1/2(z)) after a single dose of Liposome in fasting condition.

CONTACTS AND LOCATIONS:
Locations (1):
- Daniele Hamamoto, Campinas, São Paulo, Brazil